CLINICAL TRIAL: NCT04257539
Title: Influence of Reducing Sedentary Behavior on Symptoms, Inflammation and Endocannabinoids in Patients With Chronic Low Back Pain and Elevated Depressive Symptoms
Brief Title: Reducing Sedentary Time in Chronic Low Back Pain: Sedentary Intervention Using Motivational Interviewing and Technology
Acronym: SUMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Jacob Meyer, Assistant Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-068
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Chronic Low-back Pain
Keywords: Sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: The 40 participants with chronic low back pain were randomized to either Intervention or Wait-list Control groups, while all 20 healthy control participants did not receive the intervention.
Who Masked: Investigator
Masking Description: The investigator was masked to treatment group and all analyses were performed on masked data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): These subjects will participate in a behavioral intervention that will focus on reducing sedentary behavior. This will include an initial, in-person behavioral intervention with a health coach trained and a 4 week phone call. Participants will receive a wrist-worn activity prompter to aid in sedentary behavior reduction.
  Interventions: Behavioral: Intervention to Reduce Sedentary Time
- Wait-list Control Group (No Intervention): Chronic low back pain participants in this group will not receive the intervention until completion of the study. Over the 8 week intervention period, participants will be asked to maintain currently levels of physical activity, sedentary behaviors, and treatment for low back pain.
- Pain-free Control Group (No Intervention): These subjects will be healthy, pain-free adults and receive no intervention. Over the 8 week intervention period, participants in this group will be asked to maintain currently levels of physical activity, sedentary behaviors, and medication regimen.

INTERVENTIONS:
Behavioral: Intervention to Reduce Sedentary Time — Chronic low back pain participants in the intervention group will be provided with a wrist-worn activity device that vibrates after prolonged sedentariness and meet with a health coach trained in motivational interviewing to discuss individual sedentary levels and provide education surrounding sitting habits and strategies for new habit development. Participants will meet with the health coach initially and at 4 weeks during the 8 week intervention period.
  Arms: Intervention Group

SUMMARY:
This study will test the effects of a sedentary behavior intervention on pain processing, blood bio-markers and pain symptoms in individuals with chronic low back pain. The behavioral intervention will include a wrist-worn activity monitor that will notify participants when they have been sedentary for too long, motivational interviewing, and habit development.

DETAILED DESCRIPTION:
Chronic low back pain (cLBP) is a prevalent and costly condition that is associated with substantial individual and societal burden. Exercise is a recommended behavioral treatment but adherence to regular exercise is frequently low in individuals with cLBP, so research of the utility of other behavioral treatments is needed. Previous research suggests that reducing sitting time (or sedentary time) may improve symptoms of back pain and be beneficial in treating chronic low back pain. Thus, the purpose of this study is to examine the utility of a theory-based intervention to reduce sedentary time (Sedentary-intervention Utilizing Motivational Interviewing and Technology, or 'SUMIT') in individuals with cLBP. Specifically, the primary aim of this study is to examine the utility of SUMIT on sedentary behaviors in individuals with cLBP and elevated symptoms of depression. Secondary aims are to determine how SUMIT influences mood, pain symptoms, and pain psychophysics, and to quantify cytokine and endocannabinoid responses to acute exercise across the intervention. To test this, individuals with cLBP will either be randomized into an intervention group (n=20) or a wait-list control group (n=20). Additionally, healthy adults (n=20) without cLBP will be enrolled to serve as a pain-free control group and will not receive the intervention. All participants will complete baseline assessments, enroll in an 8-week intervention period, return for final assessments and a 3-month follow up. Over the intervention period, those in the intervention group will be provided with a wrist-worn activity monitor that vibrates after prolonged sedentariness and a behavioral intervention utilizing motivational interviewing and education surrounding sitting habits and strategies for new habit development. Individuals in the cLBP wait-list control group and pain-free control group will be asked to maintain current physical activity levels, sedentary behaviors, and medication and/or treatment for low back pain during this period. The investigators hypothesize that 1) objectively-monitored prolonged sedentary behavior will decrease across SUMIT and be maintained at follow-up, 2) cLBP symptoms, mood-related symptoms, and pain psychophysics (e.g pain regulation and modulation) will improve across SUMIT with maintenance of changes at follow-up, and 3) in response to acute exercise, cytokine and endocannabinoid responses post-SUMIT will become more similar to those of controls. If effective, this scalable intervention could be implemented as a behavioral treatment for cLBP.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (Currently experiencing low back pain every day or nearly every day for longer than 3 months)
* Elevated depressive symptoms (Patient Health Questionnaire-9 greater than or equal to 5)
* Ability to safely complete exercise session (Physical Activity Readiness Questionnaire)
* Willing to wear a physical activity tracker with an idle alert
* Regular access to computer or smartphone

Exclusion Criteria:

* Currently using activity tracker with idle alert
* Taking immunomodulatory medication
* Taking anti-depressant medication
* Changed medication or treatment in last 8 weeks
* Have injuries or conditions that prevent change in activity level
* Pregnant or planning to become pregnant during study enrollment

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline monitor-assessed sedentary time at 8 weeks | baseline and immediately following intervention (8 weeks)
  Average daily sedentary time in bouts longer than 60 minutes assessed using thigh worn activPAL monitors. The activPAL classifies time into sedentary, upright and stepping, has been validated for measuring free-living sedentary behaviors and is sensitive to changes in these behaviors.
Change from baseline depressive symptoms at 8 weeks | baseline, immediately following intervention (8 weeks), and 3-months after intervention
  The Patient Health Questionnaire (PHQ-9), consisting of 9 questions, will be used for participants to report the presence and severity of depressive symptoms over the past 2 weeks. PHQ-9 total score for the nine items ranges from 0 to 27. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Change from baseline low back pain symptoms at 8 weeks | baseline, immediately following intervention (8 weeks), and 3-months after intervention
  The Minimal Dataset for Low Back Pain will be used for participants to report current symptoms of low back pain and impact on daily life. On this questionnaire, for each item a score of 1 is least severe and 5 most severe, with the exception of the single item on pain intensity, which ranges from 0 (no pain) to 10 (worst possible pain). Total scores range from 8 (least impact) to 50 (most impact).
Change from baseline pain sensitivity levels at 8 weeks | before exercise at baseline and immediately following intervention (8 weeks)
  Pain sensitivity will be asesssed using the Medoc Pathway Pain & Sensory Evaluation System and applying thermal stimuli to the palm of the non-dominant hand. Subjects will be randomly presented temperatures ranging from 41°to 49°C and asked to rate each stimulus using two separate category-ratio scales to assess pain intensity and unpleasantness.
Change from baseline pain inhibition at 8 weeks | after exercise at baseline and immediately following intervention (8 weeks)
  Exercise-induced hypoalgesia (EIH) will be used to assess pain inhibition. EIH will be tested by re-administering the pain-sensitivity protocol post exercise.
Change from baseline plasma cytokine levels at 8 weeks | before and after exercise at baseline and immediately following intervention (8 weeks)
  Blood samples will be collected and processed to determine concentrations of IL-6 and TNF-alpha.
Change from baseline plasma endocannabinoid levels at 8 weeks | before and after exercise at baseline and immediately following intervention (8 weeks)
  Blood samples will be collected and processed to determine levels of anandamide(AEA) and 2-arachidonoylglycerol (2-AG).

SECONDARY OUTCOMES:
Change from baseline 36-Item Short Form Survey (SF-36) scores at 8 weeks | baseline, immediately following intervention, and 3-months after intervention
  SF-36 is a patient health and quality of life questionnaire consisting of 36 questions with the following sections: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability, so a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change from baseline Profile of Mood States Short Form scores at 8 weeks | baseline, immediately following intervention, and 3-months after intervention
  This measure asks 36 questions and assesses different dimensions of mood, including: tension, anger, vigor, fatigue, depression, and confusion. Participants rate the extent to which adjectives describe them during the past week using a 1-5 Likert scale. Totals are created for each subscale (Tension, Depression, Anger, Fatigue, Confusion, and Vigor), with higher ratings indicating greater levels of that subscale. Total Mood Disturbance is calculated by adding the first 5 subscales and then subtracting Vigor, with higher scores indicating greater mood disturbance.
Change from baseline self-reported sedentary time at 8 weeks | baseline, immediately following intervention, and 3-months after intervention
  The SIT Q 7d will be used for participants to recall their sedentary time over the past 7 days in different domains, including eating meals, transportation, occupation, screen-time, and other. Participants report levels of sitting in each domain, with higher amounts indicated great total sedentary time.
Change from baseline monitor-assessed physical activity at 8 weeks | baseline and immediately following intervention
  Average light, moderate and vigorous physical activity per day will be assessed with a thigh-worn activPAL monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No